CLINICAL TRIAL: NCT06590168
Title: Hard and Soft Tissue Changes Following Vestibular Socket Preservation Versus Ice Cream Cone Technique for Management of Defective Fresh Extraction Sockets in the Esthetic Zone: A Randomized Clinical Trial
Brief Title: Hard and Soft Tissue Changes Following Vestibular Socket Preservation Versus Ice Cream Cone Technique for Management of Defective Fresh Extraction Sockets
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nesma Mohamed Fouad Shemais, Lecturer of Periodontology, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AAN.2
Record Dates: First submitted 2024-09-03; First posted 2024-09-19 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Socket Shield; Socket Preservation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention Vestibular Socket Preservation for socket preservation (Experimental)
  Interventions: Procedure: Socket Preservation by vestibular socket therapy
- ice cream cone technique for socket preservation (Active Comparator)
  Interventions: Procedure: Socket Preservation by icecream cone technique

INTERVENTIONS:
Procedure: Socket Preservation by vestibular socket therapy — Subperiosteal tunnel will be created from the facial aspect of the socket orifice and extending apically until the extent of the vestibular access incision. A cortical shield will be introduced from the vestibular incision through the tunnel and the Socket will be filled by xenograft . Apical cut will be made at the palatal aspect to free the pedicle flap connective tissue and the pedicle flap will be raised using periosteal elevator and rotated and rolled occlusally to seal the socket and sutured using interrupted sutures . The primary palatal flap will be sutured in place over the donor site palatally using interrupted sutures.
  Arms: intervention Vestibular Socket Preservation for socket preservation
Procedure: Socket Preservation by icecream cone technique — Collagen barrier membrane will be shaped as an ice cream cone and placed in the extraction socket lining the buccal tissues. The socket will be filled with Demineralized Bovine Bone Matrix DBBM.The upper part of the membrane will be used to cover the socket and will be stabilized by interrupted sutures using prolene sutures of size 6-0
  Arms: ice cream cone technique for socket preservation

SUMMARY:
Evaluation of hard and soft tissue changes following vestibular socket preservation versus ice cream cone technique for management of defective fresh extraction sockets in the esthetic zone.

DETAILED DESCRIPTION:
The aim of this randomized clinical trial is to assess the volumetric and radiographic ridge contour changes following alveolar ridge preservation using Vestibular socket preservation in patient with type II fresh extraction sockets, versus ice cream cone technique.

In patients needing extraction in anterior maxilla with type II sockets, there will be no difference between the Vestibular socket preservation and ice cream cone technique regarding the changes in alveolar ridge contour.

ELIGIBILITY:
Inclusion Criteria:

Adults from the age of 18 - 60 years Patients with non-restorable maxillary teeth/tooth indicated for extraction in the area from 2nd premolar to 2nd premolar Type II sockets will be selected as revealed by Cone beam computed tomography (CBCT).

Intact gingival tissue with at least 2mm keratinized tissue Absence of any systemic disease or drugs that contraindicate oral surgery using Modified Cornell Medical Index . Patients accepts to provide informed consent

Exclusion Criteria:

Pregnant and lactating females. Smokers as smoking is a contraindication for any plastic periodontal surgery. Patients with BOP>15%. Patients with periodontal diseases . Handicapped and mentally retarded patients. Patients undergoing radiotherapy. Presence of systemic disease that would affect wound healing. Presence of active infection with soft tissue communication.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-07-15 (Actual); Primary Completion 2025-03-15 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Linear buccal distance (mm) | 6 months
  Soft tissue linear buccal distance will be measured using 3D scans via intaoral digital scanner at baseline, 3 months and 6 months using 3D software (NemoSmile Design 3D, Nemotec, Madrid, Spain) and STL viewer (3Shape Ortho viewer, 3Shape, Denmark)

SECONDARY OUTCOMES:
Changes in the height of the socket buccal and palatal ridges (mm) | 6 months
  Radiographic assessment using Cone Beam Computed Tomography to assess the labiopalatal alveolar ridge width reduction and changes in the height of the socket buccal and lingual ridges. Cone Beam Computed Tomography (CBCT) (Carestream Health, CS 8100 3D System) will be performed preoperative, baseline and 6 months postoperative.
Labiopalatal volumetric ridge contour analysis (mm) | 6 months
  Labiopalatal volumetric ridge contour analysis will be measured using 3D scans via intaoral digital scanner at baseline, 3 months and 6 months using 3D software (NemoSmile Design 3D, Nemotec, Madrid, Spain) and STL viewer (3Shape Ortho viewer, 3Shape, Denmark) and scans will be superimposed on each other.
Patient satisfaction (Yes/No) | 2 weeks
  Patient satisfaction will be evaluated using questionnaires during the 2 weeks after ARP.
Pain (1-10) | 2 weeks
  The severity of subjective pain and swelling will be evaluated using the visual analog scale (VAS) score (score range = 0-10, with 0 reflecting no pain and swelling), and durations of pain and swelling will be investigated during the 2 weeks after ARP

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo University, Cairo, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided